CLINICAL TRIAL: NCT05266378
Title: The Effect of Pectoralis Nerve Block on Quality of Recovery in Patients Undergoing Breast-conservative Surgery
Brief Title: Pectoralis Nerve Block and Quality of Recovery in Mastectomy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 3-2021-0468
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 1. Control arm: Conventional Anesthesia
  2. Interventional arm: Conventional Anesthesia with pectoralis nerve block.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All researchers other than the anesthesiologist who manage the randomization table and the medical staff in charge of the patient must keep the group assignment blinded until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Experimental): The group undergoing PECs block
  Interventions: Procedure: PECs block
- Control group (Placebo Comparator): The group not receiving PECs block
  Interventions: Other: Not receiving PECs Block

INTERVENTIONS:
Procedure: PECs block — The PECs block is performed immediately after induction of anesthesia, and 0.375% concentration of ropivacaine (carbiropivacaine injection, Fresinius Kavi Korea Co., Ltd.) is used with a 25 G 5 cm (or 8 cm) needle to induce ultrasound-guided pectoralis major (pectoralis major). 10mL (PECs I block) into the fascia between the pectoralis minor muscle) and the pectoralis minor muscle, and 20mL (PECs II block) between the pectoralis minor and serratus anterior muscle.
  Arms: Block group
Other: Not receiving PECs Block — In this group, the PECs block was not implemented.
  Arms: Control group

SUMMARY:
Effects of pectoralis nerve block on quality of recovery after breast surgery has been debated. We hypothesized there might exist relevant psychosocial factor or variable of pain sensitivity which would influence on the benefit of nerve block.

This study aims to assess effect of pectoralis nerve block on QoR-15 score in subgroups stratified by such factors.

DETAILED DESCRIPTION:
Study population All of patients will undergo partial mastectomy. 140 patients will be enrolled.

Intervention Pectoralis nerve block will be performed in the Block group.

Psychosocial factor screening Pain-detect, HADS, EQ-5D, PHQ-15 (somatic symptom), PCS (pain catastrophizing), BFI (big five inventory), HAM-A&D, Pressure algometry (Pain sensitivity), Quantitative sensory test (pinprick)

Study endpoints Quality of recovery (QoR)-15 Pain visual analogue scale Opioid consumption Breast Cancer Pain Questionnaire (BCPQ)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 80 years who underwent partial mastectomy for breast cancer.

Exclusion Criteria:

* Patients with a history of previous breast surgery
* Patients with a history of adverse reactions to local anesthetics
* Patients with a history of drug addiction
* Patients with cancer other than breast
* Patients with chronic pain who require analgesics
* History of hospitalization for psychiatric disorders
* Preoperative pulse oximetry (SpO2) < 95 %
* Left ventricular ejection fraction < 40%
* Moderate or severe hepatic impairment
* Body mass index over 35 kg/m2
* Blood clotting disorders
* Pregnant/lactating women
* Inability to understand consent forms and answer research questionnaires due to cognitive impairment
* Unable to read consent form (eg illiterate, foreigner, etc.)
* do not perform axillary lymph node dissection

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-02-23 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
QoR-15 | Postoperative day 1
  To compare the difference in the quality of recovery between groups, the QoR-15 questionnaire is administered on the 1st day after surgery.

SECONDARY OUTCOMES:
Intensity of pain | Postoperative day 0, 1
  Intensity of pain will be recorded by using VAS (0-10).

OTHER OUTCOMES:
Preoperative psychological factors: HADS | 1-5 days before surgery, 1st OPD visit after surgery
  Presence of anxiety and depression symptoms will be assessed by HADS (Hospital Anxiety and Depression Scale) questionnaire.
Preoperative psychological factors: EQ-5D | 1-5 days before surgery, 1st OPD visit after surgery
  Presence of anxiety and depression symptoms will be assessed by EQ-5D.
Preoperative psychological factors and pain sensitivity test: PHQ-15 | 1-5 days before surgery, 1st OPD visit after surgery
  Presence of anxiety, depression symptoms and pain sensitivity will be assessed by PHQ-15.
Preoperative psychological factors and pain sensitivity test: pain catastrophizing scale | 1-5 days before surgery, 1st OPD visit after surgery
  Presence of anxiety, depression symptoms and pain sensitivity will be assessed by pain catastrophizing scale.
Preoperative psychological factors: big five inventory | 1-5 days before surgery, 1st OPD visit after surgery
  Presence of anxiety and depression symptoms will be assessed by big five inventory.
Preoperative psychological factors: HAM-A&D | 1-5 days before surgery, 1st OPD visit after surgery
  Presence of anxiety and depression symptoms will be assessed by HAM-A&D.
Patient State Index | perioperative period
  Depth of anesthesia will be recorded by using frontal electroencephalogram (Patient State Index, The PSi is a processed EEG parameter that is related to the effect of anesthetic agents, and takes into consideration, among other factors: (1) changes in power in various EEG frequency bands; (2) changes in symmetry and synchronization between critical brain regions; and (3) the inhibition of regions of the frontal cortex.) during operation
analgesic nociception index | perioperative period
  Intensity of pain will be recorded by using analgesic nociception index during operation

CONTACTS AND LOCATIONS:
Locations (1):
- Young Song, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdallah FW, Patel V, Madjdpour C, Cil T, Brull R. Quality of recovery scores in deep serratus anterior plane block vs. sham block in ambulatory breast cancer surgery: a randomised controlled trial. Anaesthesia. 2021 Sep;76(9):1190-1197. doi: 10.1111/anae.15373. Epub 2021 Jan 25. PMID 33492696